CLINICAL TRIAL: NCT04643925
Title: Eight Weeks of Androgen Priming by hCG Before IVF/ICSI in Women With Low Ovarian Reserve
Brief Title: hCG Priming in Women With Low Ovarian Reserve
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Kristine Loessl, Consultant, PhD, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 73908
Record Dates: First submitted 2020-11-04; First posted 2020-11-25 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Infertility, Female; Ovarian Reserve; In Vitro Fertilization
Keywords: IVF; Poor ovarian reserve; Controlled ovarian stimulation; Ovarian stimulation; hCG priming
MeSH Terms: conditions — Infertility, Female | interventions — Chorionic Gonadotropin

STUDY DESIGN:
Intervention Model Description: Women will undergo two identical consecutive IVF/ICSI treatments: a Control cycle including blastocyst culture and freeze-all and a subsequent identical Study cycle, separated by eight weeks of androgen priming by daily hCG-injections. Both IVF/ICSI cycles are performed in the fixed GnRH-antagonist protocol using a daily dose of 300 IU rFSH initiated from cd 2-3 and the GnRH antagonist (Fyremadel 0.25 mg) from stimulation day 5-6.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- hCG priming (Experimental): Control cycle: A standard IVF/ICSI cycle in the fixed GnRH-antagonist protocol using a daily dose of 300 IU rFSH initiated from cd 2-3 and the GnRH antagonist (Fyremadel 0.25 mg) from stimulation day 5-6 followed by blastocyst culture and a freeze-all strategy.
  Study cycle: hCG priming by Ovitrelle 260 IE once daily for 8 weeks followed by a standard IVF/ICSI cycle in the fixed GnRH-antagonist protocol using a daily dose of 300 IU rFSH initiated from cd 2-3 and the GnRH antagonist (Fyremadel 0.25 mg) from stimulation day 5-6 followed by a single blastocyst transfer at day 5.
  Interventions: Drug: Ovitrelle

INTERVENTIONS:
Drug: Ovitrelle — Ovitrelle 260 IE once daily for 8 weeks prior to IVF/ICSI

SUMMARY:
The aim of this trial is to examine the possible effects of hCG administration for eight weeks prior to IVF/ICSI in women with low ovarian reserve. Primary outcome is the proportion of the antral follicle count that reach the pre-ovulatory stage.

DETAILED DESCRIPTION:
One of the fundamental goals in In Vitro Fertilisation (IVF) is obtaining a high number of good quality oocytes, in order to select and transfer embryos with the highest possible implantation potential thereby optimizing the chance of a pregnancy and ultimately a live birth. This is done by applying an individualized controlled ovarian stimulation (iCOS) protocol, primarily based on ovarian reserve markers like antral follicle count (AFC) and Anti-Müllerian hormone (AMH), when deciding the follicle stimulating hormone (FSH) stimulation dose. Certain patients, the so called "poor ovarian responders' (PORs), pose a clinical challenge because they have a poor ovarian reserve and develop a limited number of pre-ovulatory follicles in respond to ovarian stimulation despite high FSH stimulation doses, thus experiencing reduced live birth rates.

The aim of the present study is to examine the possible effects of long-term LH activity by the administration of hCG for eight weeks in between two identical IVF/ICSI cycles and compare cycle characteristics and outcome. The primary outcome is the follicular output rate (FORT) which reflects the proportion of antral follicles at the start of controlled ovarian stimulation that reaches the pre-ovulatory state. Secondary outcomes include amongst others AMH and antral follicle count at baseline (cd 2-3), number of pre-ovulatory follicles, oocytes retrieved, and embryos developed.

We hypothesize that eight weeks of androgen priming by hCG increases the proportion of antral follicles that reaches the pre-ovulatory state during controlled ovarian stimulation for IVF/ICSI in women with poor ovarian reserve.

ELIGIBILITY:
Inclusion Criteria:

* Regular menstrual cycle (23-35 days)
* 1.-5. IVF/ICSI cycle at inclusion
* AMH < 6.29 pmol/L (Elecsys® AMH assay)

Exclusion Criteria:

* Uterine malformations or hydrosalpinx
* Submucosal uterine myomas
* Uterine polyps
* Allergy to standard IVF/ICSI medication
* Endometriosis stage III-IV
* Severe comorbidity
* Preimplantation genetic testing
* Testicular sperm aspiration/extraction
* Tumors in the hypothalamus or pituitary gland
* Active thromboembolic disease

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2020-12-27 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Follicular output rate | Through study completion, an average of 5 months
  Follicular Output Rate (FORT: pre-ovulatory follicle count (>16 mm) at hCG trigger day/antral follicle count at baseline (2-10 mm).

SECONDARY OUTCOMES:
Antral follicle count (≤10 mm) at baseline (cd 2-3) | Through study completion, an average of 5 months
AMH at baseline (CD 2-3) | Through study completion, an average of 5 months
Number of pre-ovulatory follicles >16 mm on trigger day | Through study completion, an average of 5 months
Number of follicles >14 mm and >12 mm, >10 mm and ≤10 mm on hCG trigger day | Through study completion, an average of 5 months
Number of oocytes retrieved | Through study completion, an average of 5 months
Number of mature (MII) oocytes | Through study completion, an average of 5 months
Number of fertilized eggs (2pn) | Through study completion, an average of 5 months
Number of cleaved day 2 embryos | Through study completion, an average of 5 months
Number of good quality day 2 embryos | Through study completion, an average of 5 months
Number of top quality day 2 embryos | Through study completion, an average of 5 months
Number of blastocysts (Gardner score 1-6) | Through study completion, an average of 5 months
Number of good quality blastocysts day 5/6 | Through study completion, an average of 5 months
Number of vitrified embryos/blastocysts | Through study completion, an average of 5 months
Total number of transferred or vitrified blastocysts | Through study completion, an average of 5 months
The number of cancelled cycles and the reasons for cancellation in the two groups | Through study completion, an average of 5 months
Serum and follicular fluid hormonal levels (AMH, estradiol, progesterone, 17-OH-progesterone, hCG, LH, FSH, testosterone, androstenedione and Inhibin B | Through study completion, an average of 5 months
Granulosa/cumulus cell FSH and LH receptor expression | 1 year
Cumulus/corona gene expression analysis by quantitative PCR using three predictive genes (EFNB2, SASH1, CAMK1D). | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Anja B Pinborg, MD, Study Director — The Fertility Department, Rigshospitalet
Locations (1):
- Rigshospitalet, København Ø, Denmark

IPD SHARING:
Plan to Share IPD: Yes
On request, the study protocol and unidentifiable individual study data collected during the trial, including stored biobank samples, can be shared with research groups with relevant aims and a methodologically sound proposal. Approvals by necessary ethic committees and the Danish Data Protection Agency will be needed before sharing of data. All costs for data sharing will be covered by the party requesting the data. Data cannot be shared with groups working on research projects with the same aims, secondary aims or purposes. Furthermore, no data can be shared until 3 months after publication of first papers on the primary and secondary outcomes in this study. Biobank samples cannot be shared with research groups outside Denmark. Proposals of data sharing should be directed to anja.bisgaard.pinborg@regionh.dk. To gain access, data requestors will need to sign a data sharing agreement.
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Friis Wang N, Bogstad JW, Petersen MR, Pinborg A, Yding Andersen C, Lossl K. Androgen and inhibin B levels during ovarian stimulation before and after 8 weeks of low-dose hCG priming in women with low ovarian reserve. Hum Reprod. 2023 Sep 5;38(9):1807-1815. doi: 10.1093/humrep/dead134. PMID 37354554
- [Derived] Friis Wang N, Bogstad JW, Pors SE, Petersen MR, Pinborg A, Yding Andersen C, Lossl K. Eight weeks of androgen priming by daily low-dose hCG injections before ICSI treatment in women with low ovarian reserve. Hum Reprod. 2023 Apr 3;38(4):716-725. doi: 10.1093/humrep/dead012. PMID 36721920